CLINICAL TRIAL: NCT03801148
Title: A Phase 1, Randomized, Open-Label, Single-Center, Single-Dose, Two-Period, Two-Part Crossover Study in Healthy Subjects to Compare the Bioavailability of Dexlansoprazole From Dexlansoprazole Delayed-Release Capsules 30 mg and 60 mg Manufactured by Takeda GmbH Plant Oranienburg Relative to Dexlansoprazole Delayed-Release Capsules 30 mg and 60 mg Manufactured by Takeda Pharmaceutical Company Limited Osaka Plant Following a High-Fat Meal
Brief Title: A Study to Compare the Bioavailability (BA) of Dexlansoprazole Delayed-release Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-390MR-1002; U1111-1224-9781 (Registry Identifier: WHO)
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1:Dexlansoprazole 30mg (TOB) + Dexlansoprazole 30mg (TPC) (Experimental): Dexlansoprazole 30 mg, delayed-release capsule manufactured by TOB (Regimen A [test]), orally, once, after a high fat/calorie breakfast on Day 1 of Period 1, followed by minimum of 5 day washout period, followed by dexlansoprazole 30 mg, delayed-release capsule manufactured by TPC (Regimen B [reference]), orally, once, after a high fat/calorie breakfast on Day 1 of Period 2.
  Interventions: Drug: 30 mg dexlansoprazole capsules manufactured at TOB; Drug: 30 mg dexlansoprazole capsules manufactured at TPC
- Part 1:Dexlansoprazole 30mg (TPC) + Dexlansoprazole 30mg (TOB) (Experimental): Dexlansoprazole 30 mg, delayed-release capsule manufactured by TPC (Regimen B [reference]), orally, once, after a high fat/calorie breakfast on Day 1 of Period 1, followed by minimum of 5 day washout period, followed by dexlansoprazole 30 mg, delayed-release capsule manufactured by TOB (Regimen A [test]), orally, once, after a high fat/calorie breakfast on Day 1 of Period 2.
  Interventions: Drug: 30 mg dexlansoprazole capsules manufactured at TOB; Drug: 30 mg dexlansoprazole capsules manufactured at TPC
- Part 2:Dexlansoprazole 60mg (TOB) + Dexlansoprazole 60mg (TPC) (Experimental): Dexlansoprazole 60 mg, delayed-release capsule manufactured by TOB (Regimen C [test]), orally, once, after a high fat/calorie breakfast on Day 1 of Period 1, followed by minimum of 5 day washout period, followed by dexlansoprazole 60 mg, delayed-release capsule manufactured by TPC (Regimen D [reference]), orally, once, after a high fat/calorie breakfast on Day 1 of Period 2.
  Interventions: Drug: 60 mg dexlansoprazole capsules manufactured at TOB; Drug: 60 mg dexlansoprazole capsules manufactured at TPC
- Part 2:Dexlansoprazole 60mg (TPC) + Dexlansoprazole 60mg (TOB) (Experimental): Dexlansoprazole 60 mg, delayed-release capsule manufactured by TPC (Regimen D [reference]), orally, once, after a high fat/calorie breakfast on Day 1 of Period 1, followed by minimum of 5 day washout period, followed by dexlansoprazole 60 mg, delayed-release capsule manufactured by TOB (Regimen C [test]), orally, once, after a high fat/calorie breakfast on Day 1 of Period 2.
  Interventions: Drug: 60 mg dexlansoprazole capsules manufactured at TOB; Drug: 60 mg dexlansoprazole capsules manufactured at TPC

INTERVENTIONS:
Drug: 30 mg dexlansoprazole capsules manufactured at TOB — Dexlansoprazole delayed-release capsules.
  Arms: Part 1:Dexlansoprazole 30mg (TOB) + Dexlansoprazole 30mg (TPC); Part 1:Dexlansoprazole 30mg (TPC) + Dexlansoprazole 30mg (TOB)
Drug: 30 mg dexlansoprazole capsules manufactured at TPC — Dexlansoprazole delayed-release capsules.
  Arms: Part 1:Dexlansoprazole 30mg (TOB) + Dexlansoprazole 30mg (TPC); Part 1:Dexlansoprazole 30mg (TPC) + Dexlansoprazole 30mg (TOB)
Drug: 60 mg dexlansoprazole capsules manufactured at TOB — Dexlansoprazole delayed-release capsules.
  Arms: Part 2:Dexlansoprazole 60mg (TOB) + Dexlansoprazole 60mg (TPC); Part 2:Dexlansoprazole 60mg (TPC) + Dexlansoprazole 60mg (TOB)
Drug: 60 mg dexlansoprazole capsules manufactured at TPC — Dexlansoprazole delayed-release capsules.
  Arms: Part 2:Dexlansoprazole 60mg (TOB) + Dexlansoprazole 60mg (TPC); Part 2:Dexlansoprazole 60mg (TPC) + Dexlansoprazole 60mg (TOB)

SUMMARY:
The purpose of this study is to assess the BA of 30 or 60 milligram (mg) dexlansoprazole capsule manufactured at TOB (Takeda GmbH Plant Oranienburg) to the corresponding 30 or 60 mg dexlansoprazole manufactured at TPC (Takeda Pharmaceutical Company Ltd.).

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. Dexlansoprazole is being tested in healthy participants to compare the BA of dexlansoprazole capsules manufactured by TOB relative to dexlansoprazole capsules manufactured by TPC, under fed conditions. The study consists of two parts: Part 1 participants will receive dexlansoprazole 30 mg capsules manufactured by TOB and TPC in a crossover fashion; Part 2 participants will receive dexlansoprazole 60 mg capsules manufactured by TOB and TPC in a crossover fashion.

The study will enroll approximately 120 participants. Participants will be randomly assigned (by chance, like flipping a coin) to 1 of the 4 treatment sequences as following:

* Part 1: Dexlansoprazole 30 mg (TOB) + Dexlansoprazole 30 mg (TPC)
* Part 1: Dexlansoprazole 30 mg (TPC) + Dexlansoprazole 30 mg (TOB)
* Part 2: Dexlansoprazole 60 mg (TOB) + Dexlansoprazole 60 mg (TPC)
* Part 2: Dexlansoprazole 60 mg (TPC) + Dexlansoprazole 60 mg (TOB)

All participants will be asked to take capsule of assigned dexlansoprazole on Day 1, 30 minutes following the beginning of a high-fat/high calorie breakfast of each treatment period.

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 86 days. Participants will be contacted by phone call approximately 10 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has a body mass index (BMI) from 18 to 30 kilogram per square meter (kg/m^2), at Screening.
2. Is willing and able to consume the high-fat/high-calorie breakfast administered during the study.

Exclusion Criteria:

1. Has a history of drug abuse (defined as any illicit drug use) or drug addiction in the 12 months prior to Screening or a history of alcohol abuse (defined as regular consumption exceeding 21 units per week [1 unit equal (=) 12 ounces (oz) beer, 1.5 oz hard liquor, or 5 oz wine]) within 1 year prior to the Screening Visit, or is unwilling to agree to abstain from alcohol and drugs throughout the study.
2. Has a positive test result for drugs of abuse (defined as any illicit drug use) or alcohol at Screening or Check-in (Day -1 of Period 1).
3. Has received any known hepatic or renal clearance altering agents (example, erythromycin, cimetidine, barbiturates, phenothiazines, fluvoxamine, etc) for a period of 28 days prior to Day 1 of Period 1.
4. Has donated blood products (such as plasma) within 30 days or has donated whole blood or lost 450 milliliter (mL) or more of his or her blood volume, or had a transfusion of any blood product within 56 days prior to Day 1 of Period 1.
5. With the exception of acetaminophen, the subject has taken any excluded medication, supplements, or food products or beverages containing grapefruit or grapefruit juice, star fruit or star fruit juice, Seville-type (sour) oranges and marmalade, apple, orange, or pineapple juice, vegetables from the mustard green family (example, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard), and charbroiled meats. Hormonal contraception and hormone replacement therapy are allowed, as long as the subject has been on a stable dose for a minimum of 90 days prior to Day 1 of Period 1.
6. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch nicotine gum, e-cigarettes) within 28 days prior to Check-in (Day -1 of Period 1), or has a positive cotinine test at Screening or Check-in (Day -1 of Period 1), or is unwilling to abstain from these products for the duration of the study.
7. Has received dexlansoprazole or lansoprazole in a previous clinical study or as a therapeutic agent within 6 months of screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 10 January 2019 to 09 April 2019.
Pre-assignment Details: Healthy participants were enrolled in this 2-part and 2-way crossover study to receive dexlansoprazole 30 milligram (mg) capsules manufactured by Takeda GmbH Plant Oranienburg (TOB) and 30 mg capsules manufactured by Takeda Pharmaceutical Company Ltd. (TPC) in Part 1 and dexlansoprazole 60 mg capsules by TOB and 60 mg capsules by TPC in Part 2.
Groups:
- Part 1: Dexlansoprazole 30 mg TOB + Dexlansoprazole 30 mg TPC: Dexlansoprazole 30 mg, delayed-release capsule manufactured by TOB (test), orally, once, after a high fat/calorie breakfast on Day 1 of Period 1, followed by minimum of 5-day washout period, followed by dexlansoprazole 30 mg, delayed-release capsule manufactured by TPC (reference), orally, once, after a high fat/calorie breakfast on Day 1 of Period 2.
- Part 1: Dexlansoprazole 30 mg TPC + Dexlansoprazole 30 mg TOB: Dexlansoprazole 30 mg, delayed-release capsule manufactured by TPC (reference), orally, once, after a high fat/calorie breakfast on Day 1 of Period 1, followed by minimum of 5 day washout period, followed by dexlansoprazole 30 mg, delayed-release capsule manufactured by TOB (test), orally, once, after a high fat/calorie breakfast on Day 1 of Period 2.
- Part 2: Dexlansoprazole 60 mg TOB + Dexlansoprazole 60 mg TPC: Dexlansoprazole 60 mg, delayed-release capsule manufactured by TOB (test), orally, once, after a high fat/calorie breakfast on Day 1 of Period 1, followed by minimum of 5 day washout period, followed by dexlansoprazole 60 mg, delayed-release capsule manufactured by TPC (reference), orally, once, after a high fat/calorie breakfast on Day 1 of Period 2.
- Part 2: Dexlansoprazole 60 mg TPC + Dexlansoprazole 60 mg TOB: Dexlansoprazole 60 mg, delayed-release capsule manufactured by TPC (reference), orally, once, after a high fat/calorie breakfast on Day 1 of Period 1, followed by minimum of 5 day washout period, followed by dexlansoprazole 60 mg, delayed-release capsule manufactured by TOB (test), orally, once, after a high fat/calorie breakfast on Day 1 of Period 2.
Period: Period 1 (2 Days)
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB + Dexlansoprazole 30 mg TPC | Part 1: Dexlansoprazole 30 mg TPC + Dexlansoprazole 30 mg TOB | Part 2: Dexlansoprazole 60 mg TOB + Dexlansoprazole 60 mg TPC | Part 2: Dexlansoprazole 60 mg TPC + Dexlansoprazole 60 mg TOB
Started | 31 | 31 | 30 | 30
Completed | 30 | 30 | 30 | 30
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Period: Washout Period (at Least 5 Days)
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB + Dexlansoprazole 30 mg TPC | Part 1: Dexlansoprazole 30 mg TPC + Dexlansoprazole 30 mg TOB | Part 2: Dexlansoprazole 60 mg TOB + Dexlansoprazole 60 mg TPC | Part 2: Dexlansoprazole 60 mg TPC + Dexlansoprazole 60 mg TOB
Started | 30 | 30 | 30 | 30
Completed | 30 | 30 | 29 | 29
Not Completed | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Period 2 (2 Days)
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB + Dexlansoprazole 30 mg TPC | Part 1: Dexlansoprazole 30 mg TPC + Dexlansoprazole 30 mg TOB | Part 2: Dexlansoprazole 60 mg TOB + Dexlansoprazole 60 mg TPC | Part 2: Dexlansoprazole 60 mg TPC + Dexlansoprazole 60 mg TOB
Started | 30 | 30 | 29 | 29
Completed | 30 | 30 | 29 | 29
Not Completed | 0 | 0 | 0 | 0
Period: Follow-Up (12 Days)
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB + Dexlansoprazole 30 mg TPC | Part 1: Dexlansoprazole 30 mg TPC + Dexlansoprazole 30 mg TOB | Part 2: Dexlansoprazole 60 mg TOB + Dexlansoprazole 60 mg TPC | Part 2: Dexlansoprazole 60 mg TPC + Dexlansoprazole 60 mg TOB
Started | 30 | 30 | 29 | 29
Completed | 30 | 29 | 28 | 29
Not Completed | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who enrolled into the study and received at least one dose of the study drug(s).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB + Dexlansoprazole 30 mg TPC | Part 1: Dexlansoprazole 30 mg TPC + Dexlansoprazole 30 mg TOB | Part 2: Dexlansoprazole 60 mg TOB + Dexlansoprazole 60 mg TPC | Part 2: Dexlansoprazole 60 mg TPC + Dexlansoprazole 60 mg TOB | Total
Number analyzed (Participants) | 31 | 31 | 30 | 30 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 30 | 30 | 122
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 15 | 17 | 69
  Male | 12 | 13 | 15 | 13 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 25 | 24 | 23 | 96
  Not Hispanic or Latino | 7 | 6 | 6 | 7 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 4 | 1 | 6
  White | 30 | 29 | 25 | 27 | 111
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 31 | 30 | 30 | 122

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Dexlansoprazole
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post dose
Population: The pharmacokinetic (PK) evaluable set included all participants who enrolled into study and received at least one dose of study drug, were not discontinued from study and replaced with other participants, who completed PK sampling in both periods, complied sufficiently with protocol, and displayed evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Groups:
- Part 1: Dexlansoprazole 30 mg TOB: Dexlansoprazole 30 mg, delayed-release capsule manufactured by TOB (test), orally, once on Day 1 of Period 1 or 2.
- Part 1: Dexlansoprazole 30 mg TPC: Dexlansoprazole 30 mg, delayed-release capsule manufactured by TPC (reference), orally, once on Day 1 of Period 1 or 2.
- Part 2: Dexlansoprazole 60 mg TOB: Dexlansoprazole 60 mg, delayed-release capsule manufactured by TOB (test), orally, once on Day 1 of Period 1 or 2.
- Part 2: Dexlansoprazole 60 mg TPC: Dexlansoprazole 60 mg, delayed-release capsule manufactured by TPC (reference), orally, once on Day 1 of Period 1 or 2.
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB | Part 1: Dexlansoprazole 30 mg TPC | Part 2: Dexlansoprazole 60 mg TOB | Part 2: Dexlansoprazole 60 mg TPC
Number analyzed (Participants) | 60 | 60 | 57 | 57
nanogram/milliliter (ng/mL) | 610.1 (52.0) | 622.5 (49.9) | 1381 (45.3) | 1302 (50.3)
Statistical Analysis 1: Comparison: Part 1: Dexlansoprazole 30 mg TOB vs Part 1: Dexlansoprazole 30 mg TPC; Test type: Equivalence — Natural log (ln)-transformed-Cmax, was analyzed using an analysis of variance (ANOVA) model to assess the relative bioavailability of dexlansoprazole 30 mg capsule manufactured at TOB compared with dexlansoprazole 30 mg capsule manufactured at TPC. Geometric least square mean (LSM) ratios were calculated using the exponentiation of the difference between treatment LSM from the analyses on the ln-transformed Cmax; Geometric LSM ratio = 0.9800, 90% CI 2-sided [0.9171 to 1.0473]
Statistical Analysis 2: Comparison: Part 2: Dexlansoprazole 60 mg TOB vs Part 2: Dexlansoprazole 60 mg TPC; Test type: Equivalence — ln-transformed-Cmax, was analyzed using an ANOVA model to assess the relative bioavailability of dexlansoprazole 60 mg capsule manufactured at TOB compared with dexlansoprazole 60 mg capsule manufactured at TPC. Geometric LSM ratios were calculated using the exponentiation of the difference between treatment LSM from the analyses on the ln-transformed Cmax; Geometric LSM ratio = 1.0737, 90% CI 2-sided [1.0025 to 1.1501]

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Dexlansoprazole
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post dose
Population: The PK evaluable set included all participants who enrolled into study and received at least one dose of study drug, were not discontinued from study and replaced with other participants, who completed PK sampling in both periods, complied sufficiently with protocol, and displayed evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter(ng*hour/mL)
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB | Part 1: Dexlansoprazole 30 mg TPC | Part 2: Dexlansoprazole 60 mg TOB | Part 2: Dexlansoprazole 60 mg TPC
Number analyzed (Participants) | 60 | 60 | 57 | 57
nanogram*hour per milliliter(ng*hour/mL) | 2881 (66.8) | 2756 (62.8) | 6608 (58.5) | 6278 (59.4)
Statistical Analysis 1: Comparison: Part 1: Dexlansoprazole 30 mg TOB vs Part 1: Dexlansoprazole 30 mg TPC; Test type: Equivalence — ln-transformed- AUClast, was analyzed using an ANOVA model to assess the relative bioavailability of dexlansoprazole 30 mg capsule manufactured at TOB compared with dexlansoprazole 30 mg capsule manufactured at TPC. Geometric LSM ratios were calculated using the exponentiation of the difference between treatment LSM from the analyses on the ln-transformed AUClast; Geometric LSM ratio = 1.0455, 90% CI 2-sided [1.0070 to 1.0855]
Statistical Analysis 2: Comparison: Part 2: Dexlansoprazole 60 mg TOB vs Part 2: Dexlansoprazole 60 mg TPC; Test type: Equivalence — ln-transformed- AUClast, was analyzed using an ANOVA model to assess the relative bioavailability of dexlansoprazole 60 mg capsule manufactured at TOB compared with dexlansoprazole 60 mg capsule manufactured at TPC. Geometric LSM ratios were calculated using the exponentiation of the difference between treatment LSM from the analyses on the ln-transformed AUClast; Geometric LSM ratio = 1.0610, 90% CI 2-sided [1.0192 to 1.1046]

3. Primary Outcome: AUC0_infobs: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity Calculated Using the Observed Value of the Last Quantifiable Concentration for Dexlansoprazole
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post dose
Population: PK evaluable set: participants enrolled into study, received at least one dose of study drug, were not discontinued from study and replaced with other participants, completed PK sampling in both periods, complied sufficiently with protocol, displayed evaluable PK profiles. PK analysis population where data at specified time points was available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB | Part 1: Dexlansoprazole 30 mg TPC | Part 2: Dexlansoprazole 60 mg TOB | Part 2: Dexlansoprazole 60 mg TPC
Number analyzed (Participants) | 58 | 54 | 57 | 53
ng*hour/mL | 2927 (66.2) | 2885 (63.9) | 6734 (60.3) | 6220 (56.8)
Statistical Analysis 1: Comparison: Part 1: Dexlansoprazole 30 mg TOB vs Part 1: Dexlansoprazole 30 mg TPC; Test type: Equivalence — ln-transformed- AUC0_infobs, was analyzed using an ANOVA model to assess the relative bioavailability of dexlansoprazole 30 mg capsule manufactured at TOB compared with dexlansoprazole 30 mg capsule manufactured at TPC. Geometric LSM ratios were calculated using the exponentiation of the difference between treatment LSM from the analyses on the ln-transformed AUC0_infobs; Geometric LSM ratio = 1.0553, 90% CI 2-sided [1.0186 to 1.0933]
Statistical Analysis 2: Comparison: Part 2: Dexlansoprazole 60 mg TOB vs Part 2: Dexlansoprazole 60 mg TPC; Test type: Equivalence — ln-transformed- AUC0_infobs, was analyzed using an ANOVA model to assess the relative bioavailability of dexlansoprazole 60 mg capsule manufactured at TOB compared with dexlansoprazole 60 mg capsule manufactured at TPC. Geometric LSM ratios were calculated using the exponentiation of the difference between treatment LSM from the analyses on the ln-transformed AUC0_infobs; GMR = 1.0468, 90% CI 2-sided [1.0027 to 1.0929]

4. Primary Outcome: AUC0_infpred: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity Calculated Using the Predicted Value of the Last Quantifiable Concentration for Dexlansoprazole
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB | Part 1: Dexlansoprazole 30 mg TPC | Part 2: Dexlansoprazole 60 mg TOB | Part 2: Dexlansoprazole 60 mg TPC
Number analyzed (Participants) | 58 | 54 | 57 | 53
ng*hour/mL | 2926 (66.2) | 2884 (63.9) | 6733 (60.3) | 6217 (56.8)
Statistical Analysis 1: Comparison: Part 1: Dexlansoprazole 30 mg TOB vs Part 1: Dexlansoprazole 30 mg TPC; Test type: Equivalence — ln-transformed- AUC0_infpred, was analyzed using an ANOVA model to assess the relative bioavailability of dexlansoprazole 30 mg capsule manufactured at TOB compared with dexlansoprazole 30 mg capsule manufactured at TPC. Geometric LSM ratios were calculated using the exponentiation of the difference between treatment LSM from the analyses on the ln-transformed AUC0_infpred; Geometric LSM ratio = 1.0555, 90% CI 2-sided [1.0188 to 1.0935]
Statistical Analysis 2: Comparison: Part 2: Dexlansoprazole 60 mg TOB vs Part 2: Dexlansoprazole 60 mg TPC; Test type: Equivalence — ln-transformed- AUC0_infpred, was analyzed using an ANOVA model to assess the relative bioavailability of dexlansoprazole 60 mg capsule manufactured at TOB compared with dexlansoprazole 60 mg capsule manufactured at TPC. Geometric LSM ratios were calculated using the exponentiation of the difference between treatment LSM from the analyses on the ln-transformed AUC0_infpred; Geometric LSM ratio = 1.0472, 90% CI 2-sided [1.0029 to 1.0934]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (Day 37)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB | Part 1: Dexlansoprazole 30 mg TPC | Part 2: Dexlansoprazole 60 mg TOB | Part 2: Dexlansoprazole 60 mg TPC
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61 | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61 | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 4/61 | 3/61 | 7/59 | 5/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Dexlansoprazole 30 mg TOB (N=61) | Part 1: Dexlansoprazole 30 mg TPC (N=61) | Part 2: Dexlansoprazole 60 mg TOB (N=59) | Part 2: Dexlansoprazole 60 mg TPC (N=59)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 4 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT03801148/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT03801148/SAP_001.pdf